CLINICAL TRIAL: NCT05781334
Title: Identifying Barriers to and optiMizing In-hosPitaL usE of Evidenced-based Medical thErapies for patieNTs With Cardio-Renal-Metabolic Disease
Brief Title: Optimizing In-hospital Use of Evidence-based Therapies for Patients With Cardio-Renal-Metabolic Disease
Acronym: IMPLEMENT-CRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00112465
Record Dates: First submitted 2023-02-16; First posted 2023-03-23 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure; Type 2 Diabetes; Chronic Kidney Diseases
Keywords: heart failure; type 2 diabetes; chronic kidney disease; implementation; hospitalization
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Consult Intervention (Active Comparator): The intervention will consist of a quality improvement (QI)-based virtual consult designed by a multi-disciplinary team that will aim to address provider-level, patient-level, and system-level barriers to cardio-renal-metabolic disease medications.
  Interventions: Other: Virtual Consult Intervention
- Usual Care (No Intervention): Usual care

INTERVENTIONS:
Other: Virtual Consult Intervention — The intervention will consist of a quality improvement (QI)-based virtual consult designed by a multi-disciplinary team that will aim to address provider-level, patient-level, and system-level barriers to cardio-renal-metabolic disease medications
  Arms: Virtual Consult Intervention

SUMMARY:
This study will be a prospective randomized implementation trial for patients hospitalized with heart failure, chronic kidney disease, and/or type 2 diabetes mellitus within Duke University Medical Center. The primary hypothesis is that a virtual quality improvement-based consult intervention will improve the rate of in-hospital evidence-based cardio-renal-metabolic medication use, particularly SGLT2 inhibitor therapy. Approximately 200 patients meeting eligibility criteria will be included in the study. Patients will be assigned into study groups, as defined by randomization of their treating clinician team to receiving the virtual consult versus not.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized adults age ≥ 18 years with ≥1 of the following diagnoses, as defined by the medical record:

1. HF (any ejection fraction)
2. CKD with estimated GFR ≥ 20 mL/min/1.73m2 *
3. T2DM (by clinical history or hemoglobin A1c)

Exclusion Criteria:

1. End-stage stage renal disease on dialysis or eGFR <20 mL/kg/1.73m2.
2. Pre-menopausal woman who are either breast-feeding or pregnant
3. History of heart transplant or actively listed for heart transplant
4. Implanted left ventricular assist device or implant anticipated within 3 months.
5. Enrolled in or planning to enroll in hospice care.
6. Active cancer (except localized prostate, breast, or non-melanoma skin cancers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients prescribed SGLT2i (sodium glucose co-transporter-2 inhibitors) | hospital discharge (up to approximately 14 days)
Proportion of patients prescribed SGLT2i (sodium glucose co-transporter-2 inhibitors) | 30 days post-discharge (approximately 6 weeks)

OTHER OUTCOMES:
Number of participants with ACEI/ARB therapy among patients with heart failure or chronic kidney disease | hospital discharge (up to approximately 14 days), 30 days post-discharge (approximately 6 weeks)
Number of participants with ARNI for heart failure | hospital discharge (up to approximately 14 days), 30 days post-discharge (approximately 6 weeks)
Number of participants with Beta-blocker therapy for heart failure with ejection fraction <50% | hospital discharge (up to approximately 14 days), 30 days post-discharge (approximately 6 weeks)
Number of participants with Mineralocorticoid receptor antagonist for heart failure | hospital discharge (up to approximately 14 days), 30 days post-discharge (approximately 6 weeks)
Number of participants with GLP-1 receptor agonist for type 2 diabetes | hospital discharge (up to approximately 14 days), 30 days post-discharge (approximately 6 weeks)
Number of participants with GLP-1 receptor agonist and/or SGLT2i for type 2 diabetes | hospital discharge (up to approximately 14 days), 30 days post-discharge (approximately 6 weeks)
Composite medication score at discharge based on the use of ≥ 50% target dosing of ACEI/ARB/ARNI and beta-blocker, any MRA dose, and any SGLT2i dose (for patients with heart failure and ejection fraction </=40% only). | hospital discharge (up to approximately 14 days), 30 days post-discharge (approximately 6 weeks)
Number of participants with all-cause hospital readmission | 30 days post-discharge (approximately 6 weeks)
Number of participants with heart failure readmission | 30 days post-discharge (approximately 6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Greene, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No